CLINICAL TRIAL: NCT02395952
Title: Comparison of Standard of Care Treatments for Post-operative Non-healing Epithelial Defects
Brief Title: Healing of Persistent Epithelial Defects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Assistant Professor of Ophthalmology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001309
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Cornea
Keywords: cornea; epithelial defect; amniotic membrane
MeSH Terms: conditions — Corneal Diseases | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lubrication (Active Comparator)
  Interventions: Drug: carboxymethylcellulose sodium
- Bandage Contact Lens (Active Comparator): Acuvue Oasys Contact Lens
  Interventions: Device: Acuvue Oasys Bandage Contact Lens
- Prokera (Active Comparator): Wet amniotic membrane mounted on plastic retaining ring
  Interventions: Device: Prokera
- Ambiodisk (Active Comparator): Freeze dried amniotic membrane
  Interventions: Device: Ambiodisk

INTERVENTIONS:
Drug: carboxymethylcellulose sodium — frequent topical lubrication with artificial tears
  Arms: Lubrication
Device: Acuvue Oasys Bandage Contact Lens
  Arms: Bandage Contact Lens
Device: Ambiodisk
  Arms: Ambiodisk
Device: Prokera
  Arms: Prokera

SUMMARY:
The purpose of this study is to compare the relative efficacy of four different treatment modalities (i.e. aggressive lubrication, bandage contact lens, Ambiodisk amniotic membrane, Prokera amniotic membrane) in the healing of persistent corneal epithelial defects following retina surgery.

ELIGIBILITY:
3.1 Inclusion Criteria

* Adults aged 18 and older (inclusive) at the time of study enrollment
* Recent history of retina surgery
* Presence of persistent epithelial defect 7 days or later after surgery
* English speaking

3.2 Exclusion Criteria

* Non-English speaking patients
* Inability to incapacity to provide consent for the study
* History of corneal epithelial or limbal stem cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Abscence of persistent epithelial defect | 22 days

SECONDARY OUTCOMES:
Rate of epithelial healing in mm2/day | 22 days
Infection | 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Eye Center, Hershey, Pennsylvania, United States